CLINICAL TRIAL: NCT02116296
Title: Multifactorial Evidence Based Approach Using Behavioural Models in Understanding and Promoting Fun, Healthy Food, Play and Policy for the Prevention of Obesity in Early Childhood
Brief Title: Multi-component, Kindergarten-based, Family-involved Intervention for the Prevention of Childhood Obesity:The ToyBox-study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Yannis Manios, Associate Professor, Harokopio University
Purpose: Prevention
Other Study IDs: ToyBox-study
Record Dates: First submitted 2014-04-02; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Prevention of Childhood Obesity

ARMS (1):
- LIfestyle counseling (Other)
  Interventions: Behavioral: ToyBox-intervention

INTERVENTIONS:
Behavioral: ToyBox-intervention

SUMMARY:
The ToyBox proposal addresses Knowledge-Based Bio-Economy (KBBE)-2009-2-1-03 - Behavioural models for prevention of obesity, with a particular focus on children. It will primary aim to influence children's behaviours and prevent obesity in early childhood. The proposal will identify key behaviours related to early childhood obesity and their determinants and evaluate behavioural models and educational strategies. Based on the obtained insights at a local level, a multidisciplinary team will develop and implement a school based family involved intervention programme that could be applied on a European scale. Process, impact, outcome and cost-effectiveness evaluation will be conducted to support decision making for European Public Health Policy. The combined use of Precede-Proceed Model and Intervention Mapping will provide the framework for the development, implementation and evaluation of the ToyBox intervention. To achieve this, the project will be subdivided into 10 Work Packages (WPs). This carefully planned stepwise approach will include systematic reviews, secondary analyses of existing data sets, focus group research and school policies overview. The ToyBox project consortium spans the necessary multidisciplinary variety of experts such as public health experts, epidemiologists, nutritionists, physical activity experts, pedagogists, psychologists, behavioural scientists, nutritionists, paediatricians, early childhood psychologists, health economists, totalling 15 partners, from 10 countries. The consortium, consists of 11 universities, 1 research institute, 2 advocacy groups and a small to medium enterprise (SME) representing all regions of Europe. The consortium has ample experience in conducting and coordinating multi-centre international research as well as undertaking dissemination activities to all relevant stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 3.5 and 5 years at the time of recruitment (i.e. born between January 2007 and December 2008)
* signed consent form provided by parents/caregivers
* not participating in any other clinical trial or other health-oriented project during the academic years 2012-2013 and 2013-2014

Ages: 42 Months to 66 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-03; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Harokopio University of Athens, Kallithea, Attica, Greece

REFERENCES:
- [Derived] Flores-Barrantes P, De Miguel-Etayo P, Iglesia I, ChinAPaw MJ, Cardon G, De Craemer M, Iotova V, Usheva N, Kulaga Z, Kotowska A, Koletzko B, Birnbaum J, Manios Y, Androutsos O, Moreno LA, Gibson EL; ToyBox-study Group. Longitudinal associations between food parenting practices and dietary intake in preschool children: The ToyBox Study. Nutrition. 2024 Aug;124:112454. doi: 10.1016/j.nut.2024.112454. Epub 2024 Apr 6. PMID 38788341
- [Derived] Latomme J, Cardon G, De Bourdeaudhuij I, Iotova V, Koletzko B, Socha P, Moreno L, Androutsos O, Manios Y, De Craemer M; ToyBox-study group. Effect and process evaluation of a kindergarten-based, family-involved intervention with a randomized cluster design on sedentary behaviour in 4- to 6- year old European preschool children: The ToyBox-study. PLoS One. 2017 Apr 5;12(4):e0172730. doi: 10.1371/journal.pone.0172730. eCollection 2017. PMID 28380053
- [Derived] De Craemer M, De Decker E, Verloigne M, De Bourdeaudhuij I, Manios Y, Cardon G; ToyBox-study group. The effect of a cluster randomised control trial on objectively measured sedentary time and parental reports of time spent in sedentary activities in Belgian preschoolers: the ToyBox-study. Int J Behav Nutr Phys Act. 2016 Jan 5;13:1. doi: 10.1186/s12966-015-0325-y. PMID 26733186